CLINICAL TRIAL: NCT06492980
Title: Safety and Effectiveness of a Triple-branched Stent Graft for Arch Repair During Open Aute Debakey Type I Dissection Surgery - a Randomized Controlled Multicenter Clinical Trial
Brief Title: A Triple-branched Stent Graft for Aute Debakey Type I Dissection Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Liang-Wan Chen MD, Professor, Fujian Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A202101
Record Dates: First submitted 2023-11-08; First posted 2024-07-09 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Acute Aortic Dissection

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Triple-branched stent graft group (Experimental): The device in this clinical trial implanted covered stents in the aortic arch, three branches, and descending thoracic aorta, replacing surgical anastomosis with interventional treatment.
  Interventions: Procedure: triple-branched stent graft
- Aortic arch replacement with frozen elephant trunk (Active Comparator): This surgical method is ascending aorta + arch replacement + elephant trunk stent , that is, artificial blood vessels are used to replace the ascending aorta and aortic arch, arch anastomosis or three-branch blood vessel anastomosis is performed in the aortic arch, and a covered stent is placed in the descending thoracic aorta (Frozen Elephant Trunk Technique).
  Interventions: Procedure: triple-branched stent graft

INTERVENTIONS:
Procedure: triple-branched stent graft — a triple-branched stent graft for aortic arch repairement during surgery

SUMMARY:
Prospective, multicenter, randomized controlled clinical trial plan to evaluate the effectiveness and safety of intraoperative stent system in the treatment of acute type I aortic dissection

DETAILED DESCRIPTION:
Acute aortic dissection is a local rupture in the aortic intima. Blood flows into the middle layer from the rupture, causing the middle layer of the aortic wall to tear along the long axis, tearing the complete aortic wall into the dissected intima (intima + part of the middle layer) and the dissected outer wall (part of the middle layer + outer layer), and forming a true lumen (the original aortic lumen) and a false lumen (the cavity between the dissected intima and the dissected outer wall). The torn dissected outer wall bears the pressure of the entire aorta, which can easily cause aortic rupture. The clinical characteristics of this disease are acute onset and rapid progression, making it one of the most dangerous and fatal cardiovascular diseases. Acute type I aortic dissection involves the ascending aorta, aortic arch and the entire aorta, and is the most dangerous type of acute aortic dissection. At present, surgery is the only treatment for acute type I aortic dissection.

Since the most common rupture site of acute aortic dissection is in the ascending aorta, clinical trials have shown that simple ascending aortic replacement can effectively save the lives of most patients with acute type I aortic dissection, and this operation is simple and suitable for emergency rescue of such critically ill patients. Therefore, simple ascending aortic replacement has become a classic emergency surgical method for acute type I aortic dissection.

However, most patients with acute type I aortic dissection after simple ascending aortic replacement have residual false lumens in the aortic arch and its distal aorta (i.e., dissection lesions still exist). The expansion and rupture of these residual false lumens are the most important factors affecting the long-term efficacy after surgery.

During the operation, reconstruction of the aortic arch as much as possible, elimination of the intimal rupture of the arch and the proximal descending aorta, expansion of the true lumen, and promotion of thrombosis in the false lumen are the fundamental ways to improve the long-term effect after surgery. Therefore, for patients with a high probability of residual false lumen expansion and rupture, such as young patients, patients with a long postoperative survival time, and patients with multiple ruptures in the aortic arch, most scholars currently advocate that the aortic arch should be reconstructed at the same time as the ascending aorta replacement, and the four-branch artificial blood vessel is often used to replace the aortic arch, and the descending aorta fixed elephant trunk technique (Frozen Elephant Trunk Technique) is an effective method for the treatment of acute aortic dissection developed in recent years. It can effectively close the aortic intimal rupture, promote thrombosis in the false lumen, and expand the true lumen. In order to simplify the reconstruction of the aortic arch in acute type I aortic dissection, we designed an integrated three-branch covered stent system (referred to as the intraoperative stent system), which is implanted under direct vision during surgery to repair the aortic arch, that is, the three-branch covered stent is sent into the arch, the root of the branch artery and the descending part of the arch under deep hypothermic circulatory arrest to cover the rupture of the dissection in the arch, the root of the branch artery and the descending part of the arch, and the proximal end of the stent and the distal incision of the ascending aorta are directly anastomosed with the artificial blood vessel replacing the ascending aorta. This avoids the anastomosis of the three branches of the aortic arch, reduces the difficulty of surgery, and shortens the time of cerebral ischemia and lower body ischemia.

This clinical trial adopts a prospective, multicenter, randomized controlled method, with the marketed product descending aortic elephant trunk stent implantation (Frozen Elephant Trunk Technique) as a control, and evaluates the effectiveness and safety of the intraoperative stent system as a test device in the treatment of acute type I aortic dissection through a standardized experimental design.

This experimental device is an upgraded product of Beijing Yuhengjia Technology Co., Ltd.'s existing products. It was developed by Beijing Yuhengjia Technology Co., Ltd. and has transferred a full set of technical documents to Yuhengjia (Xiamen) Technology Co., Ltd.

Beijing Yuhengjia Technology Co., Ltd. uses the same materials and the same process to produce similar products "endovascular covered stent" for the treatment of thoracic descending aorta and abdominal aorta lesions. It has been approved by the National Medical Products Administration, obtained a product registration certificate, and used in clinical treatment, achieving the expected treatment purpose.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with acute type I aortic dissection who need arch repair;
2. Aged ≥20 years and ≤65 years;
3. Acute phase, with onset within 14 days before surgery;
4. Subjects who can understand the purpose of the trial, voluntarily participate and sign the informed consent form, and are willing to accept follow-up.

Exclusion Criteria:

1. The presence of anatomical variations, such as aortic arch malformation, aortic coarctation; common origin of the innominate artery and the left common carotid artery, aberrant right subclavian artery, abnormal origin of the left conical artery, stenosis or distortion of the branch arteries; and the diameter of the aortic arch and branch artery diameters do not match the specifications of the test device;
2. Dissection is secondary to a history of aortic treatment, Marfan syndrome, etc.
3. Aortic lesions and branch artery lesions caused by acute type I aortic dissection, including aortic pre-rupture, branch artery rupture, branch artery occlusion, and severe ischemic complications caused by poor organ perfusion, such as myocardial ischemia, stroke (ischemic brain injury), paraplegia (spinal artery ischemia), mesenteric artery ischemia, renal artery dysplasia, etc.
4. Severe infectious lesions that are not controlled;
5. Patients who need to receive other concomitant treatments, such as severe hypertension, chronic obstructive pulmonary disease, coronary heart disease, chronic kidney disease and other serious underlying lesions that require long-term treatment;
6. Patients with other life-threatening lesions, such as advanced malignant tumors, and whose expected survival time is less than one year;
7. Patients with other lesions in the heart and aorta (patients with other heart diseases that require concurrent heart surgery, such as coronary heart disease, mitral valve disease, tricuspid valve disease, etc.), who are not suitable for stent interventional treatment, such as peripheral vascular disease and blood disease;
8. Subjects who have participated in other drug or device clinical trials and have not reached the primary study endpoint; and pregnant women.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-10-27 (Actual); Primary Completion 2024-10-10 (Estimated); Study Completion 2025-10-10 (Estimated)

PRIMARY OUTCOMES:
Mortality within 30days post-operation | 30 days
  Mortality within 30days post-operation

SECONDARY OUTCOMES:
Aortic dissection-related death occurred within 12 months after surgery | 12 month
  Aortic dissection-related death occurred within 12 months after surgery
Thrombosis of the false lumen of the arch and proximal descending aorta | 12 month
  Thrombosis of the false lumen of the arch and proximal descending aorta
Technical success | 12 month
  Successful insertion, successful positioning, and patency of the lumen were used as indicators

CONTACTS AND LOCATIONS:
Overall Officials: Liang-wan Chen, M.D Ph.D, Study Chair — Fujian Medical University Union Hospital
Locations (1):
- Department of Cardiovascular Surgery, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No